CLINICAL TRIAL: NCT03528577
Title: A Randomized, Single-Dose, Double-Blind, Double-Dummy, Four-Period, Four-Sequence, Four-Treatment, Placebo and Active Controlled, Comparative, Multiple-Center, Crossover-Design, Bronchoprovocation Study to Evaluate the Pharmacodynamic Equivalence of Albuterol Sulfate Inhalation Aerosol, eq 90 mcg Base (Sun Pharmaceuticals Industries Limited) to PROAIR® HFA (Albuterol Sulfate) Inhalation Aerosol, eq 90 mcg Base (Teva Respiratory, LLC) in Subjects With Stable, Mild Asthma
Brief Title: A Study to Evaluate the Effect of of Albuterol Sulfate Inhalation Aerosol, eq 90 mcg Base (Sun Pharmaceuticals Industries Limited)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLR_17_08
Record Dates: First submitted 2018-04-21; First posted 2018-05-18 (Actual); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Test (Experimental): Albuterol Sulfate Inhalation Aerosol, eq 90 mcg
  Interventions: Drug: Zero-dose; Drug: 90 mcg of PROAIR® HFA; Drug: 180 mcg of 90 mcg of PROAIR® HFA; Drug: 90 mcg of albuterol sulfate inhalation aerosol
- Reference (Active Comparator): PROAIR® HFA (albuterol sulfate) Inhalation Aerosol, eq 90 mcg
  Interventions: Drug: Zero-dose; Drug: 90 mcg of PROAIR® HFA; Drug: 180 mcg of 90 mcg of PROAIR® HFA; Drug: 90 mcg of albuterol sulfate inhalation aerosol
- Test Placebo (Placebo Comparator): Placebo for Albuterol Sulfate Inhalation Aerosol
  Interventions: Drug: Zero-dose; Drug: 90 mcg of PROAIR® HFA; Drug: 180 mcg of 90 mcg of PROAIR® HFA; Drug: 90 mcg of albuterol sulfate inhalation aerosol
- Reference Placebo (Placebo Comparator): Placebo for Albuterol Sulfate Inhalation Aerosol
  Interventions: Drug: Zero-dose; Drug: 90 mcg of PROAIR® HFA; Drug: 180 mcg of 90 mcg of PROAIR® HFA; Drug: 90 mcg of albuterol sulfate inhalation aerosol

INTERVENTIONS:
Drug: Zero-dose — Treatment A
Drug: 90 mcg of PROAIR® HFA — Treatment B
Drug: 180 mcg of 90 mcg of PROAIR® HFA — Treatment C
Drug: 90 mcg of albuterol sulfate inhalation aerosol — Treatment D

SUMMARY:
To Evaluate the Pharmacodynamic Equivalence of Albuterol Sulfate Inhalation Aerosol, eq 90 mcg base (Sun Pharmaceuticals Industries Limited) to PROAIR® HFA (albuterol sulfate) Inhalation Aerosol, eq 90 mcg base (Teva Respiratory, LLC) in Subjects With Stable, Mild Asthma

ELIGIBILITY:
Inclusion Criteria:

1. Men or non-pregnant women 18 to 65 years of age.
2. Signed informed consent form that meets all criteria of current Food and Drug Administration (FDA) regulations.
3. Females of childbearing potential must not be pregnant or lactating (as confirmed by a negative urine pregnancy test
4. Ability to use inhalation aerosol correctly.

Exclusion Criteria:

1. Any clinically significant finding on physical exam in the opinion of the Investigator, would compromise subject's safety or data integrity.
2. Employees of the Investigator or research center or their immediate family members.
3. Previous participation in this study.
4. Inability to understand the requirements of the study and the relative information and are unable or not willing to comply with the study protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2018-09-22 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-08-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - SPARC Site 02, Miami Lakes, Florida
  - SPARC site 01, Bethesda, Maryland
  - SPARC Site 04, St Louis, Missouri
  - SPARC Site 06, Gastonia, North Carolina
  - SPARC Site 05, Edmond, Oklahoma
  - SPARC Site 07, Warwick, Rhode Island
  - SPARC Site 08, Boerne, Texas
  - SPARC Site 03, Waco, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Treatments were administered according to a four-treatment, four-period, four-sequence design.
  124 eligible subjects were randomized to each one of the four sequences: ABCD
  Sequence
  Sequence 1 : A B C D Sequence 2: D C B A Sequence 3: C A D B Sequence 4: B D A C
Groups:
- Total: Treatment A: Zero-dose : Two different Reference Placebo inhalers and two different Test Placebo inhalers
  Treatment B: 90 mcg of Reference : One Reference inhaler, one Reference Placebo inhaler, and two different Test Placebo inhalers
  Treatment C: 180 mcg of Reference Two different Reference inhalers and two different Test Placebo inhalers
  Treatment D: 90 mcg of Test One Test inhaler, one Test Placebo inhaler, and two different Reference Placebo inhalers
Period: Sequence 1
Arm/Group | Total
Started (128 subjects with persistent bronchial asthma were randomized during the study.) | 128
Completed | 126 (Per report, 119 completed the trial, and all 119 received Treatment A, B, C and D.)
Not Completed | 2
Not completed — Failed Spirometry | 1
Not completed — Restricted medication | 1
Period: Sequence 2
Arm/Group | Total
Started | 128
Completed | 125
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Failed Spirometry | 1
Period: Sequence 3
Arm/Group | Total
Started | 128
Completed | 127
Not Completed | 1
Not completed — Failed Spirometry | 1
Period: Sequence 4
Arm/Group | Total
Started | 128
Completed | 125
Not Completed | 3
Not completed — Failed Spirometry | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall Baseline: Summary of Demographic Data and Baseline Characteristics (Safety Population)
Arm/Group | Overall Baseline
Number analyzed (Participants) | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 32
  White | 96
  More than one race | 0
  Unknown or Not Reported | 0
Tobacco Use [Count of Participants; unit: Participants] | 0
Number of years patient has suffered from symptoms caused by asthma [Mean (Standard Deviation); unit: years] | 23.62 (13.17)
FEV1 (Pre-saline) [Mean (Standard Deviation); unit: Litre] — FEV1 is Forced Expiratory Volume (flow rate) in 1 second
  Litre | 3.20 (0.72)
FEV1 (Post-saline) [Mean (Standard Deviation); unit: Litre] — FEV1 is Forced Expiratory Volume (flow rate) in 1 second
  Litre | 3.23 (0.74)
PC20 FEV1 [Mean (Standard Deviation); unit: mg/mL] — PC20 is Provocative concentration (mg/mL) of methacholine required to reduce FEV1 by 20%
  FEV1 is Forced Expiratory Volume (flow rate) in 1 second
  mg/mL | 0.95 (1.36)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacodynamic Endpoint Post-dose PC20
Description: The primary pharmacodynamic endpoint is the post-dose PC20, which is the provocative concentration of methacholine challenge agent required to reduce the forced expiry volume in one second (FEV1) by 20%, following the administration of different doses of albuterol (or placebo) by inhalation.
  Primary analysis group -pharmacodynamic population.
Time Frame: Approximately 15 minutes after last inhalation of study product
Population: The statistical analysis was performed based on the Dose-Scale approach. This approach was referenced in FDA's draft Guidance on albuterol sulfate metered/inhalation and described in FDA's draft Guidance on Orlistat capsule. The PC20 data from various treatments (such as placebo, 90 mcg Test, 90 mcg Reference and 180 mcg Reference) from different study period was pooled to perform the Dose-Scale model using NONMEM. Therefore, per test arm values were not reported.
Measure: Mean (90% Confidence Interval); unit: mg/mL
Groups:
- Primary Analysis Group: This group included all randomized subjects who:
  1. completed at least 1 of the 4 randomized treatment periods with an evaluable PC20FEV1.
  2. were compliant with study treatment dosing procedures.
  3. did not use any restricted concomitant medications.
  4. did not have any other significant protocol deviations.
Arm/Group | Primary Analysis Group
Number analyzed (Participants) | 126
mg/mL | 114 [52.8 to 162.0]

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: It is the approximate duration over which adverse event data were collected
Groups:
- Treatment A: Zero-dose
- Treatment B: 90 mcg of Reference (PROAIR® HFA)
- Treatment C: 180 mcg of Reference (PROAIR® HFA)
- Treatment D: 90 mcg of Test (Albuterol Sulfate HFA Inhalation Aerosol)
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
All-Cause Mortality (participants affected / at risk) | 0/125 | 0/125 | 0/123 | 0/126
Serious Adverse Events (participants affected / at risk) | 0/125 | 0/125 | 0/123 | 0/126
Other Adverse Events (participants affected / at risk) | 7/125 | 3/125 | 9/123 | 5/126
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=125) | Treatment B (N=125) | Treatment C (N=123) | Treatment D (N=126)
influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
FEV1/FVC ratio (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
tension headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
accelerated hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-12-21): https://cdn.clinicaltrials.gov/large-docs/77/NCT03528577/SAP_001.pdf
  • Study Protocol (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/77/NCT03528577/Prot_002.pdf